CLINICAL TRIAL: NCT05254119
Title: REGISTRY PLATFORM INTO DIAGNOSIS, TREATMENT AND OUTCOME OF LUNG CANCER PATIENTS
Brief Title: DIAGNOSIS, TREATMENT AND OUTCOME OF LUNG CANCER PATIENTS
Acronym: REGISTURK-LUNG
Status: Active, not recruiting | Type: Observational
Sponsor: Mahmut Gumus (Network)
Responsible Party: Sponsor-Investigator, Mahmut Gumus, Board Member of Oncological Clinical Research Association, Oncological Clinical Research Association, Turkey
Organization: Oncological Clinical Research Association, Turkey (Network)
Other Study IDs: LUNG-RWD-001
Record Dates: First submitted 2022-02-10; First posted 2022-02-24 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Non Small Cell Lung Cancer; Small-cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; Small Cell Lung Cancer; Immunotherapy; Progression free Survival; Survival
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational, prospective clinical research, multi-center clinical research platform with the main objective to assess molecular biomarker testing, treatment and outcome of patients with NSCLC or SCLC in Turkey

DETAILED DESCRIPTION:
In Turkey, non-small cell lung cancer (NSCLC) is the most common cause of cancer-related death in men and one of the most common causes of cancer-related deaths in women. Because of the heterogeneity of NSCLC or SCLC, it is crucial to characterize the biology of the tumor as exact as possible, to predict the course of disease as accurate as possible, and to determine the optimal therapeutic algorithm as early as possible after initial diagnostic work-up.

These efforts are an obligatory part of the initial diagnostics, since thorough knowledge of the biology of the disease and the resulting therapeutic options ensure optimal care of Volunteers with NSCLC or SCLC. The aim of REGISTURK is to set up a national clinical research platform to document molecular testing, treatment and course of disease of patients with NSCLC or SCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Patient histopathologically diagnosed with non-small cell lung cancer or small cell lung cancer
2. Written informed consent no later than six weeks after start of first-line treatment
3. Age ≥ 18 years

Exclusion Criteria:

* Volunteers participating in a research program for non-small cell or small cell lung cancer that includes interventions outside of routine clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Six thousands REGISTURK patients treated at 42 study sites (university hospitals, education and research hospitals and private hospital-based oncology practices).REGISTURK sites will be selected in accordance with patients load, hospital type and geographical distribution. All patients diagnosed with NSCLC or SCLC at selected centers will be enrolled consecutively throughout the study period. All patients diagnosed with lung cancer who receive treatment or who are followed with the best supportive care approach or refuse treatment will be recorded. All approaches in this regard will be determined and the reasons will be examined. Adult male and female patients with non-small cell (early, locally advanced or metastatic) or small cell will be considered "REGISTURK-LUNG patients"
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Frequency of molecular/mutational analysis | throughout of treatment, 36 months
  To collect data on the frequency of molecular/mutational biomarker testing
Type of molecular/mutational analysis | throughout of treatment, 36 months
  To collect data on the type of molecular/mutational biomarker testing

SECONDARY OUTCOMES:
Type of treatment | throughout of treatment, 36 months
  To describe systemic treatments and sequential treatments applied in real-life practice.
The Rate of Response Rate | throughout of treatment, 36 months
  Response rate
Progression free survival time | throughout of treatment, 36 months
  Progression free survival
Overall survival time | throughout of treatment, 36 months
  Overall survival
The frequency of comorbidities | throughout of treatment, 36 months
  Comorbidities rate
Advers events rate | throughout of treatment, 36 months
  Advers events

CONTACTS AND LOCATIONS:
Locations (39):
- Turkey (Türkiye) (39):
  - Adana Başkent University Hospital, Adana
  - Adana City Training and Research Hospital, Adana
  - Ankara City Hospital (1), Ankara
  - Ankara City Hospital (2), Ankara
  - Ankara Dr. Abdurrahman Yurtaslan Oncology Training and Research Hospital, Ankara
  - Ankara Gülhane Traning and Research Hospital, Ankara
  - Ankara Liv Hospital, Ankara
  - Ankara Memorial Hospital, Ankara
  - Dıskapı Yıldırım Beyazid Training and Research Hospital, Ankara
  - Antalya Training and Research Hospital, Antalya
  - Bursa Uludağ University Hospital, Bursa
  - Canakkale 18 Mart University Medicine Faculty Hopsital, Çanakkale
  - Dicle University Medicine Faculty Hospital, Diyarbakır
  - Trakya University Medicine Faculty Hospital, Edirne
  - Erzurum Atatürk University Medicine Faculty Hospital, Erzurum
  - Gaziantep University Medicine Faculty Hospital, Gaziantep
  - Acibadem University Hospital, Istanbul
  - Akdeniz University Medicine Faculty Hospital, Istanbul
  - Bakırköy Dr. Sadi Konuk Training and Research Hospital, Istanbul
  - Bezmialem Vakıf University Hospital, Istanbul
  - Istanbul Medeniyet University, Istanbul
  - Istanbul Oncology Hospital, Istanbul
  - Istanbul Umraniye Training and Research Hsopital, Istanbul
  - Istanbul University Cerrahpasa Medicine Faculty Hospital, Istanbul
  - Kartal Dr. Lütfi Kırdar Training and Research Hospital, Istanbul
  - Marmara University Hospital, Istanbul
  - Medipol University Hospital, Istanbul
  - Pendik Medical Park Hospital, Istanbul
  - Prof.Dr. Cemil Taşcıoğlu City Hospital, Istanbul
  - Sureyyapasa Chest Disease Hospital, Istanbul
  - Ege University Medicine Fculty Hospital, Izmir
  - Izmir Medical Park Hospital, Izmir
  - Kocaeli University Hospital, İzmit
  - Erciyes Üniversity Medicine Faculty Hospital, Kayseri
  - Necmettin Erbakan University Meram Medicine Faculty Hospital, Konya
  - Inonu Uniersity Medicine Faculty Hospital, Malatya
  - Sakarya University Training and Research Hospital, Sakarya
  - Samsun Ondokuz Mayıs University Medicine Faculty Hospital, Samsun
  - Karadeniz Technical University Medicine Faculty Hospital, Trabzon

IPD SHARING:
Plan to Share IPD: Undecided